CLINICAL TRIAL: NCT03721549
Title: Evaluation of Infectivity and Illness of Norwalk GI.1 Virus Lot 001-09NV in the Human Challenge Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: WCCT Global (Industry)
Collaborators: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VXA-G11-201.1
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Norovirus Infection
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Intervention Model Description: A total of 16 eligible healthy young adults will be challenged with either the moderate or higher dose of norovirus inoculum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Dose Inoculum (Experimental): Moderate dose of Norwalk GI.1 Virus, 3.6x10^5 genome copies
  Interventions: Biological: Norwalk GI.1 Virus
- Higher Dose Inoculum (Experimental): Higher dose of Norwalk GI.1 Virus, 1x10^6 genome copies
  Interventions: Biological: Norwalk GI.1 Virus

INTERVENTIONS:
Biological: Norwalk GI.1 Virus — Norwalk virus causes viral gastroenteritis, which is also known as acute nonbacterial gastroenteritis, food poisoning, food infection, or stomach flu.

SUMMARY:
There is a need for safe, highly infectious Norovirus inocula for use in Norovirus vaccine-challenge studies to assess the efficacy of Norovirus vaccines and examine the immune response among vaccinated and unvaccinated subjects. The purpose of this study is to generate the infection and illness rate and immune response data necessary for the conduct of future investigation of Norovirus vaccine studies.

ELIGIBILITY:
Inclusion Criteria:

* General good health, without significant medical illness, based on medical history, physical examination, vital signs, and clinical laboratories (CBC, chemistry, and urinalysis) as determined by the investigator in consultation with the research monitor and sponsor
* Available for all planned visits and to spend at least 5 days in confinement
* Confirmed blood type (A or O)
* Demonstrated to be H type-1 antigen secretor positive (by saliva test)
* Body mass index between 17 and 30 at screening
* Female subjects must have a negative pregnancy test and either use contraceptives or be sterile
* Available to return for follow-up visits following discharge from the inpatient unit and deliver stool specimens to the investigator promptly

Exclusion Criteria:

* Presence of significant medical condition
* Donation or use of blood or blood products within 4 weeks prior to challenge
* Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic
* Abnormal stool pattern
* Any gastroenteritis within the past 2 weeks
* Occupational hazards, including having daily contact with children under the age of 5, women known to be pregnant, employment in the food service industry, health care workers, etc.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Costa Mesa, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Dose Inoculum | Higher Dose Inoculum
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Dose Inoculum | Higher Dose Inoculum | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.50 (6.57) | 39.88 (7.34) | 36.19 (7.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 4 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 6 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 4 | 2 | 6
  Caucasian | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 16
Secretor Status [Count of Participants; unit: Participants] — H type-1 antigen secretor positive
  Participants | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Norovirus Gastroenteritis (NVG)
Description: Occurrence of NVG within 7 days post-challenge
Time Frame: 7 days post-challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Dose Inoculum | Higher Dose Inoculum
Number analyzed (Participants) | 8 | 8
Participants | 5 | 4

2. Secondary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: Occurrence of SAEs
Time Frame: 42 ± 3 days post-challenge
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Dose Inoculum | Higher Dose Inoculum
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 45 ± 3
Arm/Group | Moderate Dose Inoculum | Higher Dose Inoculum
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Dose Inoculum (N=8) | Higher Dose Inoculum (N=8)
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03721549/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03721549/SAP_001.pdf